CLINICAL TRIAL: NCT01935986
Title: The Effect of a Probiotic on Protection Against Upper Respiratory Tract Infections in Children
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to bankruptcy of the CRO company
Sponsor: Probi AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: U-12-032
Record Dates: First submitted 2013-08-28; First posted 2013-09-05 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-01

CONDITIONS: Upper Respiratory Tract Infection
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- probiotic (Experimental): dietary supplement
  Interventions: Dietary Supplement: probiotic
- placebo (Placebo Comparator): dietary supplement without probiotic
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: probiotic
  Arms: probiotic
Dietary Supplement: placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to study the effect of a probiotic on protection against upper respiratory tract infections (URTI) in children.

ELIGIBILITY:
Inclusion Criteria:

* healthy children

Exclusion Criteria:

-

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 131 (Actual)
Dates: Start 2013-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
upper respiratory tract infections | study period, 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Foodfiles Sweden Ab, Uppsala, Sweden